CLINICAL TRIAL: NCT05317585
Title: Continuous Glucose Monitor Use and Perinatal Outcomes Among Pregnant Women With Type 2 Diabetes Mellitus: A Randomized Controlled Trial
Brief Title: Continuous Glucose Monitor Use in Pregnancy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Gianna Wilkie, Clinical Fellow in Maternal Fetal Medicine, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00001802
Record Dates: First submitted 2022-03-29; First posted 2022-04-08 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Type 2 Diabetes Treated With Insulin; Pregnancy, High Risk
Keywords: Type 2 diabetes; Pregnancy
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: This is a prospective, single center, randomized study evaluating pregnancy glycemic monitoring strategies between women with continuous glucose monitors and standard of care fingerstick glucose monitoring.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Continuous Glucose Monitoring (CGM) (Experimental): Patients will be randomized to application of a continuous glucose monitor (CGM). They will apply the device in the clinical setting and be instructed how to download their information onto their smartphones or using the CGM device reader. They will use the CGM for the duration of the pregnancy until delivery.
  Interventions: Device: Continuous Glucose Monitor
- Fingerstick Glucose Monitoring (Active Comparator): Patients will be randomized to checking their blood glucose with fingerstick monitors at time of fasting in the AM, and 2 hours after each meal. This is the standard of care for patients in the pregnancy diabetes clinic.
  Interventions: Device: Routine Capillary Blood Glucose Monitoring (Fingerstick Glucose)

INTERVENTIONS:
Device: Continuous Glucose Monitor — Continuous Glucose Monitor
  Arms: Continuous Glucose Monitoring (CGM)
Device: Routine Capillary Blood Glucose Monitoring (Fingerstick Glucose) — Routine Capillary Blood Glucose Monitoring (Fingerstick Glucose)
  Arms: Fingerstick Glucose Monitoring

SUMMARY:
The purpose of this study is to perform a randomized controlled trial among 180 pregnant women with type 2 diabetes mellitus (T2DM) comparing continuous glucose monitor (CGM) use to the standard of care of multiple daily fingerstick glucose monitoring and its impact on large for gestational age infants, maternal glycemic control, patient satisfaction, and additional adverse perinatal outcomes.

DETAILED DESCRIPTION:
A continuous glucose monitor (CGM) can provide detailed insight into daily glucose fluctuations and individual glucose patterns, and it is advised for patients with type 1 diabetes mellitus and advanced type 2 diabetes mellitus (T2DM). Despite this recommendation, pregnant women are not receiving the same standard of care. It has been studied minimally in pregnant women with T2DM, despite preliminary studies showing improvement in adverse perinatal outcomes and glycemic control among pregnant women with type 1 diabetes. Therefore, there is a paucity of data regarding CGM use among pregnant women with T2DM, and significant potential to reduce the significant multigenerational effects associated with diabetes in pregnancy with this technology.

The study team therefore propose to perform a randomized controlled trial among 180 pregnant women with T2DM comparing CGM use to the standard of care of multiple daily fingerstick glucose monitoring and its impact on large for gestational age infants, maternal glycemic control, patient satisfaction, and additional adverse perinatal outcomes.

ELIGIBILITY:
Inclusion Criteria: Women will be deemed eligible for the study by the following inclusion criteria:

* 1) age greater than or equal to 18 years old
* 2) singleton gestation less than or equal to 14 weeks at initial obstetric visit
* 3) established diagnosis of T2DM by laboratory criteria including hemoglobin A1c ≥6.5%, oral glucose tolerance test ≥200 mg/dL, or fasting plasma glucose ≥126 mg/dL
* 4) receiving prenatal care at UMASS Memorial Health Care (UMMHC) and plans to deliver at UMMHC
* 5) able and willing to provide informed consent

Exclusion Criteria: Women will be deemed ineligible for the study based on the following exclusion criteria:

* 1) known diagnosis of type 1 diabetes or gestational diabetes
* 2) plan to receive prenatal care or delivery outside of UMMHC
* 3) inability to provide informed consent
* 4) multifetal gestation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-05-23 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Large for Gestational Age Infant | Within 2 hours of birth
  The neonatal birthweight will be used to calculate large for gestational age size based on the gestational age at delivery.

SECONDARY OUTCOMES:
Third Trimester Hemoglobin A1c | Between 28 weeks and delivery
  Third Trimester Hemoglobin A1c
Mode of Delivery | At delivery
  Mode of delivery (vaginal versus cesarean)
Hypertensive Disorders of Pregnancy | After 20 weeks of gestation until delivery
  Development of gestational hypertension or pre-eclampsia after 20 weeks of gestation
Preterm Birth | At delivery
  Preterm birth (delivery less than 37 weeks gestation)
Number of participants with a shoulder dystocia | At delivery
  Number of participants with a shoulder dystocia
Neonatal Intensive Care Unit Admission (NICU) | At delivery and within first 2 days of life
  Neonatal Intensive Care Unit Admission (NICU)
Neonatal Respiratory Distress | At delivery
  Neonatal Respiratory Distress requiring respiratory support
APGAR less than 7 at 5 minutes of life | 5 Minutes after Delivery
  APGAR score less than 7 at 5 minutes of life
Number of participants with neonatal hypoglycemia | Within 2 hours of birth
  Number of participants with neonatal hypoglycemia as defined by first neonatal blood sugar obtained within 2 hours of birth
Gestational age at delivery | At Delivery
  Gestational age at delivery
Maternal Patient Satisfaction Survey with Glucose Monitoring | postpartum day 1 after delivery
  This will be assessed by the glucose monitoring satisfaction survey (GMSS) version 2. Participants will complete the survey, which contains 4 subscales and a total score. The subscales assess openness, emotional burden, behavioral burden, and worthwhileness. The higher the score the greater the satisfaction, with a total maximum score 75.

CONTACTS AND LOCATIONS:
Overall Officials: Gianna L Wilkie, MD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts Memorial Medical Center, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Feig DS, Donovan LE, Corcoy R, Murphy KE, Amiel SA, Hunt KF, Asztalos E, Barrett JFR, Sanchez JJ, de Leiva A, Hod M, Jovanovic L, Keely E, McManus R, Hutton EK, Meek CL, Stewart ZA, Wysocki T, O'Brien R, Ruedy K, Kollman C, Tomlinson G, Murphy HR; CONCEPTT Collaborative Group. Continuous glucose monitoring in pregnant women with type 1 diabetes (CONCEPTT): a multicentre international randomised controlled trial. Lancet. 2017 Nov 25;390(10110):2347-2359. doi: 10.1016/S0140-6736(17)32400-5. Epub 2017 Sep 15. PMID 28923465
- [Background] Voormolen DN, DeVries JH, Sanson RME, Heringa MP, de Valk HW, Kok M, van Loon AJ, Hoogenberg K, Bekedam DJ, Brouwer TCB, Porath M, Erdtsieck RJ, NijBijvank B, Kip H, van der Heijden OWH, Elving LD, Hermsen BB, Potter van Loon BJ, Rijnders RJP, Jansen HJ, Langenveld J, Akerboom BMC, Kiewiet RM, Naaktgeboren CA, Mol BWJ, Franx A, Evers IM. Continuous glucose monitoring during diabetic pregnancy (GlucoMOMS): A multicentre randomized controlled trial. Diabetes Obes Metab. 2018 Aug;20(8):1894-1902. doi: 10.1111/dom.13310. Epub 2018 May 8. PMID 29603547
- [Background] Secher AL, Ringholm L, Andersen HU, Damm P, Mathiesen ER. The effect of real-time continuous glucose monitoring in pregnant women with diabetes: a randomized controlled trial. Diabetes Care. 2013 Jul;36(7):1877-83. doi: 10.2337/dc12-2360. Epub 2013 Jan 24. PMID 23349548
- [Background] Murphy HR, Rayman G, Lewis K, Kelly S, Johal B, Duffield K, Fowler D, Campbell PJ, Temple RC. Effectiveness of continuous glucose monitoring in pregnant women with diabetes: randomised clinical trial. BMJ. 2008 Sep 25;337:a1680. doi: 10.1136/bmj.a1680. PMID 18818254